CLINICAL TRIAL: NCT03874104
Title: An Evaluation of the Tolerance and Acceptability of a Whey-based Extensively Hydrolysed Feed With Pre- and Probiotics, for the Dietary Management of Cows' Milk Allergy in Infants
Brief Title: Synbiotic Extensively Hydrolysed Feed Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PEPSYN001 V6
Record Dates: First submitted 2018-11-23; First posted 2019-03-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study product (Experimental): Extensively Hydrolysed Formula containing Pre- and Probiotics
  Interventions: Dietary Supplement: Extensively Hydrolysed Formula containing Pre- & Probiotics

INTERVENTIONS:
Dietary Supplement: Extensively Hydrolysed Formula containing Pre- & Probiotics — Extensively Hydrolysed Formula containing Pre- and Probiotics

SUMMARY:
This study of the tolerance and acceptability of a extensively hydrolysed formula (eHF) containing pre- and probiotics will assess gastrointestinal (GI) tolerance, product intake and acceptability in 40 infants (aged <13 months) currently using or requiring an extensively hydrolysed formula for the dietary management of CMA. Patients already prescribed an eHF (or other appropriate feed for CMA) at time of recruitment will undertake a 3 day baseline period in which their current symptoms, compliance, GI tolerance and acceptability towards their current feed is assessed, before introducing the study product for a period of 4 weeks. Patients who are not on an eHF (or other appropriate feed for CMA) at baseline will forgo this 3 day baseline period and immediately introduce the study product for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged <13 months
* Currently using or requiring an extensively hydrolysed formula for the dietary management of cows' milk allergy
* Expected to receive at least 25% of their energy intake from the study feed
* Already fed with infant formula or hypoallergenic formula (either partially or fully)
* Written, informed consent from parent/carer

Exclusion Criteria:

* "Severe" cows' milk allergy (clinically judged to require an amino acid formula) or any other contraindications to the use of an extensively hydrolysed formula
* Exclusively breastfed infants
* Primary lactose intolerance
* History of poor tolerance to whey based EHFs
* Immunocompromised infants
* Premature infants (born <37 weeks)
* Major hepatic or renal dysfunction
* Requirement for any parenteral nutrition
* Tube-fed via a post-pyloric route
* Participation in other clinical intervention studies within 1 month of recruitment to this study
* Investigator concern around the ability of family to comply with protocol and requirements of study

Max Age: 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal tolerance from baseline to intervention day 28: questionnaire | 31 days
  Gastro-intestinal tolerance will be recorded by the parent on Baseline Days 1-3 (where this period is undertaken by the patient) and on Intervention Days 1, 2, 3, 7, 14, 21, 26, 27, and 28. Tolerance will be recorded using a standardised gastro-intestinal tolerance questionnaire, to be completed by the parents/carer

SECONDARY OUTCOMES:
Compliance | 31 days
  Compliance with feed prescription will be assessed daily throughout the study by recording how much feed was received. The amount prescribed by the Dietitian will be recorded at the start of the study, and any changes to this prescription also noted. During the baseline period (where this is undertaken) the compliance of the patient's usual feed will be assessed.
Parent-reported Atopic Symptoms | 31 days
  Recorded via visual analogue scales at baseline and at the end of each week. Parents will record on a 100mm line the severity of a number of common atopic symtpoms, with the scale running from "not at all/none" at 0mm and "as bad as possible/
Food Allergy QOL - Parental burden questionnaire | 31 days
  Measured at baseline and at the end of study via a Food Allergy QOL - Parental Burden Questionnaire
Formula acceptability: Likert-style questionnaire | 31 days
  Feed acceptability will be assessed on Baseline Day 3 (for current feed, where applicable) and on the final day of the intervention period (Intervention day 28) via a Likert-style questionnaire
Nutrient intake | 31 days
  Nutrient intake, including the intake of all nutrition provided (including the study product, any other enteral tube feeding, foods, drinks etc.) will be recorded via a 24hr dietary recall, conducted by the Dietitian at the Baseline Visit and at the End of Study Visit.
Atopic dermatitis severity | 31 days
  Measured via Patient Orientated SCORing Atopic Dermatitis (PO-SCORAD) tool at Baseline, Intervention Day 7 and the final dat of the study
Change in weight | 31 days
  Weight will be measured at the start and end of the study in kg
Safety (Adverse Events) | 31 days
  Adverse events captured throughout entire study
Change in length (cm) | 31 days
  Length will be measured at the start and end of the study
Change in head circumference (cm) | 31 days
  Head circumference will be measured at the start and end of the study

CONTACTS AND LOCATIONS:
Locations (8):
- United Kingdom (8):
  - Brighton and Sussex University Hospital NHS Foundation Trust, Brighton
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Ashford and St Peter's Hospital NHS Foundation Trust, Chertsey
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Rotherham NHS Foundation Trust, Rotherham
  - university Hospitals Southampton NHS Foundation Trust, Southampton
  - West Hertfordshire NHS Foundation Trust, Watford

IPD SHARING:
Plan to Share IPD: No